CLINICAL TRIAL: NCT02682979
Title: Continuity of the Therapeutic Limitation Code: Analysis of the Variables of Admission in the Emergency Service That Are Associated With a Therapeutic Limitation Upon Exit
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Murielle Surquin, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-Therapeutic limitations
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Geriatrics
Keywords: therapeutic limitation code; emergency unit admittance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Geriatric patients: 100 consecutive geriatric patients admitted in the Emergency Department of the Brugmann Hospital, Horta site, from 01/04/2015.
  Interventions: Other: Medical files analysis

INTERVENTIONS:
Other: Medical files analysis — Retrospective analysis of the medical files according to medical, social and geriatric criteria.

SUMMARY:
Demographically, the geriatric population is expanding. It is also increasingly found in the emergency services.However, emergency services are not designed to accommodate these patients, whose needs are specific. This population is defined by complex physical and psychosocial needs, included in a comprehensive geriatric assessment too complex to be carried out in the emergency services.

Many publications focused on ways to prevent potentially avoidable visits to geriatric patients in emergency services. People rely upon a therapeutic limitation code established for these patients to determine the intensity of the care that may be given to them. However, few geriatric patients arriving in the emergency services were already given such a code.

As a consequence, the intensity of the care given to these emergency patients is influenced by the perception of the functional and cognitive status of the patient, even if part of this perception is incorrect. Moreover, it is also well established that the outcome of geriatric patients with severe pathologies at admission is often poor and that there is a need to find alternatives to the intensive treatment offered.

The goal of this study will be to determine the prevalence of the presence of a therapeutic limitation code in geriatric patients at hospital admission / admission to the emergency department, and when they leave the hospital. This will be carried out for all geriatric patients residing or placed in nursing homes at the end of the hospitalization.The investigators postulate that establishing a therapeutic limitation code for these fragile patients, before they leave the hospital for a nursing home, would reduce the number of future admissions of these patients in the emergency department.

DETAILED DESCRIPTION:
Demographically, the geriatric population is expanding. It is also increasingly found in the emergency services.However, emergency services are not designed to accommodate these patients, whose needs are specific. This population is defined by complex physical and psychosocial needs, included in a comprehensive geriatric assessment too complex to be carried out in the emergency services. The multidisciplinary care they need takes time.

Several options are investigated worldwide to properly manage these fragile patients:

* Scales of frailty and functional decline screening
* Specialized care units: the Mobile Geriatric Team, the Emergency short-stay units, the acute care geriatric unit, the geriatric nurse liaison model, or a service specific geriatric emergency.

Many publications focused on ways to prevent potentially avoidable visits to geriatric patients in emergency services. People rely upon a therapeutic limitation code established for these patients to determine the intensity of the care that may be given to them. However, few geriatric patients arriving in the emergency services were already given such a code.

As a consequence, the intensity of the care given to these emergency patients is influenced by the perception of the functional and cognitive status of the patient, even if part of this perception is incorrect. Moreover, it is also well established that the outcome of geriatric patients with severe pathologies at admission is often poor and that there is a need to find alternatives to the intensive treatment offered.

The goal of this study will be to determine the prevalence of the presence of a therapeutic limitation code in geriatric patients at hospital admission / admission to the emergency department, and when they leave the hospital. This will be carried out for all geriatric patients residing or placed in nursing homes at the end of the hospitalization.The investigators postulate that establishing a therapeutic limitation code for these fragile patients, before they leave the hospital for a nursing home, would reduce the number of future admissions of these patients in the emergency department.

Furthermore, this study offers the prospective to establish in the future a systematic implementation of the therapeutic limitation code for geriatric patients residing in nursing homes, therefore anticipating the various issues specific to his population in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the hospital via the emergency department and placed in a nursing home upon hospital discharge
* Patients will an available global geriatric evaluation (either realized in the geriatric ward, either realized by the geriatric team)

Exclusion Criteria:

* if multiple hospitalizations occur during the study length, data related to the first hospitalization only will be analyzed.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 100 consecutive geriatric patients admitted in the emergency department of the Brugmann Hospital, Horta site, from 01/04/2015 till 11/02/2016.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of a therapeutic limitation code (hospital admittance) | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  The medical files of the patients admitted in the emergency department of the hospital, from 01/04/2015, will be examined in order to determine if they had a therapeutic limitation code upon admittance.
Prevalence of a therapeutic limitation code (hospital discharge) | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  The medical files of the patients admitted in the emergency department of the hospital, from 01/04/2015, will be examined in order to determine if received a therapeutic limitation code upon hospital discharge.

SECONDARY OUTCOMES:
social status | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files. The investigators will evaluate if the social status of the patient is linked to a therapeutic limitation decision upon hospital discharge.
autonomy status | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if the autonomy of the patient is linked to a therapeutic limitation decision upon hospital discharge. Patient autonomy is evaluated by the results of either of these two tests: the Sherpa test or the Katz scale.
cognitive status | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if the cognitive status of the patient is linked to a therapeutic limitation decision upon hospital discharge. The patient cognitive status is evaluated by the results of either the confusion assessment method or the mini mental state evaluation test.
diagnosis | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if the admission motive/established diagnosis is linked to a therapeutic limitation decision upon hospital discharge.
hospitalisation length | Patients hopitalized from 01/04/2015 till present date (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if the hospitalisation length is linked to a therapeutic limitation decision upon hospital discharge.
Albumine | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if the nutrition status (albumine measurement) is linked to a therapeutic limitation decision upon hospital discharge.
Hydratation level | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if the hydration level (combined sodium and creatinine/urea measurement) is linked to a therapeutic limitation decision upon hospital discharge.
Unintentional weigh loss | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if an unintentional weigh loss is linked to a therapeutic limitation decision upon hospital discharge.
Presence of comorbidities | Patients hospitalized from 01/04/2015 till 11/02/2016 (11 months)
  Retrospective analysis of patient medical files.The investigators will evaluate if the presence of comorbidities (dementia or severe cardiac decompensation or cancer or pneumonia or severe cardio-vascular diseases or hepatic insufficiency) is linked to a therapeutic limitation decision upon hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Murielle Surquin, MD, Principal Investigator — CHU Brugmann; Axelle Gregory, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Folstein MF, Robins LN, Helzer JE. The Mini-Mental State Examination. Arch Gen Psychiatry. 1983 Jul;40(7):812. doi: 10.1001/archpsyc.1983.01790060110016. No abstract available. PMID 6860082
- [Background] Yesavage JA. Geriatric Depression Scale. Psychopharmacol Bull. 1988;24(4):709-11. No abstract available. PMID 3249773
- [Background] Clement JP, Nassif RF, Leger JM, Marchan F. [Development and contribution to the validation of a brief French version of the Yesavage Geriatric Depression Scale]. Encephale. 1997 Mar-Apr;23(2):91-9. French. PMID 9264935
- [Background] Goring H, Baldwin R, Marriott A, Pratt H, Roberts C. Validation of short screening tests for depression and cognitive impairment in older medically ill inpatients. Int J Geriatr Psychiatry. 2004 May;19(5):465-71. doi: 10.1002/gps.1115. PMID 15156548
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Katz S. Assessing self-maintenance: activities of daily living, mobility, and instrumental activities of daily living. J Am Geriatr Soc. 1983 Dec;31(12):721-7. doi: 10.1111/j.1532-5415.1983.tb03391.x. PMID 6418786
- [Background] Katz PR, Karuza J, Kolassa J, Hutson A. Medical practice with nursing home residents: results from the National Physician Professional Activities Census. J Am Geriatr Soc. 1997 Aug;45(8):911-7. doi: 10.1111/j.1532-5415.1997.tb02958.x. PMID 9256840
- [Background] Katz PP, Yelin EH. Activity loss and the onset of depressive symptoms: do some activities matter more than others? Arthritis Rheum. 2001 May;44(5):1194-202. doi: 10.1002/1529-0131(200105)44:53.0.CO;2-6. PMID 11352254
- [Background] Katz PP, Morris A. Use of accommodations for valued life activities: prevalence and effects on disability scores. Arthritis Rheum. 2007 Jun 15;57(5):730-7. doi: 10.1002/art.22765. PMID 17530671
- [Background] Derouesne C, Poitreneau J, Hugonot L, Kalafat M, Dubois B, Laurent B. [Mini-Mental State Examination:a useful method for the evaluation of the cognitive status of patients by the clinician. Consensual French version]. Presse Med. 1999 Jun 12;28(21):1141-8. French. PMID 10399508